CLINICAL TRIAL: NCT01935908
Title: Pilot Study of Seizure Prophylaxis With Levetiracetam in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Seizure Prophylaxis With Levetiracetam in Aneurysmal Subarachnoid Hemorrhage - Pilot Study
Acronym: SPLASH - Pilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SPLASH-P1
Record Dates: First submitted 2013-04-21; First posted 2013-09-05 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Subarachnoid Hemorrhage; Seizures
Keywords: Subarachnoid Hemorrhage; Seizures; Prophylaxis; Levetiracetam
MeSH Terms: conditions — Subarachnoid Hemorrhage; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): The control group will not receive levetiracetam as seizure prophylaxis.
- Treatment Group (Active Comparator): levetiracetam 500mg in adults, twice daily, administered by mouth, per tube, or IV. The route of administration will be dependent upon the patient's clinical status and ability to tolerate each form. In descending order of preference, route of administration will be: oral, per tube, IV.
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam
  Other Names: keppra
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to determine the feasibility of prospectively enrolling and randomizing patients with aneurysmal subarachnoid hemorrhage (aSAH) to receive levetiracetam or not to receive levetiracetam, and documenting in-hospital and follow-up clinical variables.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ≤ 75 years of age
* Newly diagnosed aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

* One or more antiepileptic medication is taken as a pre-admission medication
* Seizure occurrence in the field or in the emergency department, or anytime before consent could be obtained
* Inability to obtain informed consent from the patient, or from the patient's appropriate surrogate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Randomization Yield | 6 months
  The primary outcome will be the number of patients randomized to either levetiracetam administration or no administration of levetiracetam divided by the total number of aneurysmal subarachnoid hemorrhage patients who present to the Vanderbilt University Emergency Department or are directly admitted to the Neuro Intensive Care Unit. (Unit of Measure: numeric fraction)

SECONDARY OUTCOMES:
Protocol Adherence Yield | 9 months
  The Protocol Adherence Yield is calculated by dividing the number of patients completing the study without incurring a protocol deviation by the total number of patients randomized. (Unit of Measure: numeric fraction)

OTHER OUTCOMES:
modified Rankin Scale (mRS) | hospital discharge, 1-month, 3-months
  mRS - modified Rankin Scale (0-6): 0 - no symptoms
  1. - no significant disability. Able to carry out all usual activities, despite some symptoms
  2. - slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities
  3. - moderate disability. Requires some help, but able to walk unassisted.
  4. - moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - dead
Glasgow Outcomes Scale-Extended (GOSE) | hospital discharge, 1-month, 3-month
  GOSE - Glasgow Outcomes Scale - Extended (1-8):
  1. - death
  2. - vegetative state
  3. - lower severe disability
  4. - upper severe disability
  5. - lower moderate disability
  6. - upper moderate disability
  7. - lower good recovery
  8. - upper good recovery

CONTACTS AND LOCATIONS:
Overall Officials: J D Mocco, MS, MD, Principal Investigator — Vanderbilt University; Michael C Dewan, MD, Study Director — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Butzkueven H, Evans AH, Pitman A, Leopold C, Jolley DJ, Kaye AH, Kilpatrick CJ, Davis SM. Onset seizures independently predict poor outcome after subarachnoid hemorrhage. Neurology. 2000 Nov 14;55(9):1315-20. doi: 10.1212/wnl.55.9.1315. PMID 11087774
- [Background] Choi KS, Chun HJ, Yi HJ, Ko Y, Kim YS, Kim JM. Seizures and Epilepsy following Aneurysmal Subarachnoid Hemorrhage : Incidence and Risk Factors. J Korean Neurosurg Soc. 2009 Aug;46(2):93-8. doi: 10.3340/jkns.2009.46.2.93. Epub 2009 Aug 31. PMID 19763209
- [Background] Connolly ES Jr, Rabinstein AA, Carhuapoma JR, Derdeyn CP, Dion J, Higashida RT, Hoh BL, Kirkness CJ, Naidech AM, Ogilvy CS, Patel AB, Thompson BG, Vespa P; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology. Guidelines for the management of aneurysmal subarachnoid hemorrhage: a guideline for healthcare professionals from the American Heart Association/american Stroke Association. Stroke. 2012 Jun;43(6):1711-37. doi: 10.1161/STR.0b013e3182587839. Epub 2012 May 3. PMID 22556195
- [Background] Hart RG, Byer JA, Slaughter JR, Hewett JE, Easton JD. Occurrence and implications of seizures in subarachnoid hemorrhage due to ruptured intracranial aneurysms. Neurosurgery. 1981 Apr;8(4):417-21. doi: 10.1227/00006123-198104000-00002. PMID 7242892
- [Background] Hovinga CA. Levetiracetam: a novel antiepileptic drug. Pharmacotherapy. 2001 Nov;21(11):1375-88. doi: 10.1592/phco.21.17.1375.34432. PMID 11714211
- [Background] Kvam DA, Loftus CM, Copeland B, Quest DO. Seizures during the immediate postoperative period. Neurosurgery. 1983 Jan;12(1):14-7. doi: 10.1227/00006123-198301000-00003. PMID 6828220
- [Background] Lin CL, Dumont AS, Lieu AS, Yen CP, Hwang SL, Kwan AL, Kassell NF, Howng SL. Characterization of perioperative seizures and epilepsy following aneurysmal subarachnoid hemorrhage. J Neurosurg. 2003 Dec;99(6):978-85. doi: 10.3171/jns.2003.99.6.0978. PMID 14705724
- [Background] Little AS, Kerrigan JF, McDougall CG, Zabramski JM, Albuquerque FC, Nakaji P, Spetzler RF. Nonconvulsive status epilepticus in patients suffering spontaneous subarachnoid hemorrhage. J Neurosurg. 2007 May;106(5):805-11. doi: 10.3171/jns.2007.106.5.805. PMID 17542523
- [Background] Mink S, Muroi C, Seule M, Bjeljac M, Keller E. Levetiracetam compared to valproic acid: plasma concentration levels, adverse effects and interactions in aneurysmal subarachnoid hemorrhage. Clin Neurol Neurosurg. 2011 Oct;113(8):644-8. doi: 10.1016/j.clineuro.2011.05.007. Epub 2011 Jun 23. PMID 21703756
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655
- [Background] Murphy-Human T, Welch E, Zipfel G, Diringer MN, Dhar R. Comparison of short-duration levetiracetam with extended-course phenytoin for seizure prophylaxis after subarachnoid hemorrhage. World Neurosurg. 2011 Feb;75(2):269-74. doi: 10.1016/j.wneu.2010.09.002. PMID 21492729
- [Background] Beeton AG, Upton PM, Shipton EA. The case for patient-controlled analgesia. Inter-patient variation in postoperative analgesic requirements. S Afr J Surg. 1992 Mar;30(1):5-6. PMID 1566203
- [Background] Rhoney DH, Tipps LB, Murry KR, Basham MC, Michael DB, Coplin WM. Anticonvulsant prophylaxis and timing of seizures after aneurysmal subarachnoid hemorrhage. Neurology. 2000 Jul 25;55(2):258-65. doi: 10.1212/wnl.55.2.258. PMID 10908901
- [Background] Rosengart AJ, Huo JD, Tolentino J, Novakovic RL, Frank JI, Goldenberg FD, Macdonald RL. Outcome in patients with subarachnoid hemorrhage treated with antiepileptic drugs. J Neurosurg. 2007 Aug;107(2):253-60. doi: 10.3171/JNS-07/08/0253. PMID 17695377
- [Background] Shah D, Husain AM. Utility of levetiracetam in patients with subarachnoid hemorrhage. Seizure. 2009 Dec;18(10):676-9. doi: 10.1016/j.seizure.2009.09.003. Epub 2009 Oct 27. PMID 19864168
- [Background] Sundaram MB, Chow F. Seizures associated with spontaneous subarachnoid hemorrhage. Can J Neurol Sci. 1986 Aug;13(3):229-31. doi: 10.1017/s0317167100036325. PMID 3742338
- [Background] Szaflarski JP, Sangha KS, Lindsell CJ, Shutter LA. Prospective, randomized, single-blinded comparative trial of intravenous levetiracetam versus phenytoin for seizure prophylaxis. Neurocrit Care. 2010 Apr;12(2):165-72. doi: 10.1007/s12028-009-9304-y. PMID 19898966
- [Background] Usami K, Saito N. Prophylactic anticonvulsants after subarachnoid hemorrhage. World Neurosurg. 2011 Feb;75(2):214. doi: 10.1016/j.wneu.2010.09.035. No abstract available. PMID 21492717